CLINICAL TRIAL: NCT00001005
Title: Interleukin-2 Augmentation of Specific Anti-HIV Immune Responses: Phase I Trial of the Combination of 3'-Azido-3'-Deoxythymidine (Zidovudine) and Recombinant Interleukin-2 in Patients With Asymptomatic HIV Infection Associated With Lymphadenopathy (Walter Reed Stage II)
Brief Title: A Study of Zidovudine Plus Interleukin-2 in HIV-Infected Patients Who Have No Symptoms of Infection But Who Have Tender Lymph Nodes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 042; 11017 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; HIV Seropositivity; Interleukin-2; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; HIV Seropositivity; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; aldesleukin

INTERVENTIONS:
Drug: Zidovudine
Drug: Aldesleukin

SUMMARY:
AMENDED: To investigate whether subcutaneous (SC) injection of IL-2 produces biological responses which parallel those observed with IV dosing. Original design: To evaluate the short-term effects of combined administration of zidovudine (AZT) and increasing doses of recombinant interleukin-2 (aldesleukin; IL-2) in patients infected with HIV, who have lymphadenopathy, but who are otherwise asymptomatic (no other symptoms). The first phase of this clinical trial will establish maximum tolerated dose ( MTD ). How quickly the drugs get into the blood and how long they remain there (pharmacokinetics) will also be studied at each dose as well as the effect on HIV.

Since AZT has no effect on cells that contain inactive virus (latently infected cells) and these cells may act as viral reservoirs, that a second agent that can destroy these infected cells would be useful in combination with AZT. The different activities of AZT and IL-2, as well as the non-overlapping nature of their mechanisms of action and toxicity, increase the theoretical benefits of combining AZT, a drug which has clinically significant activity in HIV-related disease but cannot eliminate infected cells, with IL-2, a drug which may enhance anti-HIV immunity, destroy chronically infected cells, and allow immune recognition of latently infected cells.

DETAILED DESCRIPTION:
Since AZT has no effect on cells that contain inactive virus (latently infected cells) and these cells may act as viral reservoirs, that a second agent that can destroy these infected cells would be useful in combination with AZT. The different activities of AZT and IL-2, as well as the non-overlapping nature of their mechanisms of action and toxicity, increase the theoretical benefits of combining AZT, a drug which has clinically significant activity in HIV-related disease but cannot eliminate infected cells, with IL-2, a drug which may enhance anti-HIV immunity, destroy chronically infected cells, and allow immune recognition of latently infected cells.

Five patients who have already received and tolerated oral AZT for at least 8 weeks continue their AZT treatment and at the same time receive IL-2 on a schedule of 5 days on the drug, 2 days off the drug. The IL-2 is administered by 30-minute intravenous (IV) infusion according to this schedule for 4 weeks. The first week of IL-2 treatment is on an inpatient basis and the remaining 3 weeks are on an outpatient basis. Toxicity is monitored every week. Maximum tolerated dose (MTD) is defined as the maximum dose at which 3 out of 5 patients experience Grade 3 or above toxicity during the course of IL-2 administration. A second cohort of five patients will receive IV IL-2. If the MTD is not reached, five additional patients will receive IV IL-2. All five patients in a given cohort must complete a full 4-week course of IL-2 before subsequent patients are entered at the next higher dose level. After IV dosing is completed at these three levels, additional 5-patient cohorts receive subcutaneous (SC) IL-2 according to the same schedule. Each patient is restricted to one dosage group. Patients are treated and followed for a total of 24 weeks. Patients receive ibuprofen for fever and chills.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Necessary topical agents, including nystatin or clotrimazole, as well as acyclovir. Patients on medications without which the patient would be placed at significant risk (seizures, diabetic control, respiratory embarrassment) may continue only at the discretion of the study pharmacologist.

Patients must have:

* Asymptomatic HIV infection associated with lymphadenopathy.
* Walter Reed Stage II disease, with positive antibody to HIV confirmed by Western blot test.

Exclusion Criteria

Co-existing Condition:

Patients will be excluded from the study for the following:

* Development of a disease requiring a drug which might potentiate toxicity of the study drugs or a drug likely to have antiretroviral effect.
* Active opportunistic infection.
* Major organ allograft.
* Significant cardiac or pulmonary disease or central nervous system (CNS) lesions.

Concurrent Medication:

Excluded:

* Ongoing therapy for an opportunistic infection.
* Beta-blockers.
* Antihypertensive medication other than diuretics.
* All nonessential medication including pain medications.

Patients without interleukin 2 (IL-2) augmentable anti-HIV antibody-dependent cellular cytotoxicity (ADCC) or or cell-mediated cytotoxicity (CMC) in vitro are excluded.

Prior Medication:

Excluded within 12 weeks of study entry:

* Other antiretroviral agents (patients with CD4 counts of 400 - 500 per mm3 who are receiving AZT may continue to receive it until study treatment is initiated).
* Immunomodulators.
* Corticosteroids.
* Other experimental therapy.
* Antineoplastic chemotherapy.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Weinhold, Study Chair
Locations (1):
- Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina, United States

REFERENCES:
- [Background] Weinhold K, Tyler D, Austin A, Lyerly K, Bolognesi D, Bartlett J. Augmentation of non-mhc restricted cellular cytotoxicities in patients receiving Zidovudine plus interleukin 2. Int Conf AIDS. 1989 Jun 4-9;5:406 (abstract no WBP330)
- [Background] Bartlett JA, Blankenship KD, Greenberg M, Tyler DS, Weinhold KJ. The safety of Zidovudine and interleukin 2 in asymptomatic HIV infected patients. Int Conf AIDS. 1989 Jun 4-9;5:406 (abstract no WBP325)
- [Background] Bartlett JA, Berend C, Petroni GR, Ottinger J, Tyler DL, Pettinelli C, Weinhold KJ. Coadministration of zidovudine and interleukin-2 increases absolute CD4 cells in subjects with Walter Reed stage 2 human immunodeficiency virus infection: results of ACTG protocol 042. J Infect Dis. 1998 Oct;178(4):1170-3. doi: 10.1086/515677. PMID 9806053